CLINICAL TRIAL: NCT06169163
Title: Volatile Organic Compounds as Breath Biomarkers in Squamous Oesophageal Neoplasms
Acronym: ViSON
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Velindre NHS Trust (Other Government); Cardiff and Vale University Health Board (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Bedfordshire Hospitals NHS Foundation Trust (Other); University Hospitals, Leicester (Other); The Clatterbridge Cancer Centre NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); University Hospital Plymouth NHS Trust (Other); NHS Tayside (Other Government); NHS Highlands (Other); The Christie NHS Foundation Trust (Other); North Cumbria University Hospitals NHS Trust (Other); Maidstone & Tunbridge Wells NHS Trust (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 23SM8534
Record Dates: First submitted 2023-11-24; First posted 2023-12-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Oesophageal Squamous Cell Carcinoma; Oesophageal Cancer
Keywords: Breath biomarker; Early detection; Oesophageal cancer; Oesophageal squamous cell cancer; Volatile organic compounds
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSCC group: Patients with histopathology confirmed, treatment naive OSCC
  Interventions: Other: Exhaled breath sampling
- Non-cancer controls: Patients who are undergoing an endoscopy for non-specific upper gastrointestinal (GI) symptoms and are shown to have either:
  1. A healthy upper GI tract
  2. Benign upper gastrointestinal disease
  Interventions: Other: Exhaled breath sampling

INTERVENTIONS:
Other: Exhaled breath sampling — Participants will maintain a clear fluid diet for a minimum of 6 hours prior to breath collection. Participants will be asked to provide a breath sample by exhaling into single-use breath collection bags. Using a custom designed gas sampling pump, the breath VOCs will be transferred onto TD tubes at a controlled flow rate. This breath sampling procedure will be repeated once. When the participants' breath sampling is complete, room air (Blank) samples must be taken onto additional TD tubes using the same procedure. The TD tubes will be sealed with long-term storage caps using the CapLok Tool.

SUMMARY:
Oesophageal Squamous Cell Carcinoma (OSCC) is a cancer of the food pipe that affects around 2000 patients in the UK every year. It is often detected at an advanced stage, resulting in poor survival (5-year survival less than 20%). Early detection can improve survival (5-year survival >70%). Therefore, early detection is vital to improving survival.

There are no national screening guidelines, and an endoscopy (A camera test to look at the food pipe) is the only available test to detect OSCC.

Early detection of OSCC is challenging for many reasons. Firstly, early disease symptoms are non-specific, which patients often overlook. Secondly, 'Alarm' symptoms such as weight loss, difficulty swallowing or vomiting blood are signs of advanced stage. Lastly, endoscopy is an invasive test with associated risks and significant discomfort.

The investigators propose to develop a breath test for patients with non-specific symptoms. Breath testing has the ideal characteristics for a triage test because it is non-invasive, simple to perform, cost-effective and highly acceptable to patients. The test is based on identifying volatile organic compounds (VOCs, small molecules) that are produced by the cancer and released in breath.

The breath test will be offered by General Practitioners (GPs) to patients with non-specific symptoms. Those who test positive will be referred for an urgent camera test, and those who test negative can be reassured.

DETAILED DESCRIPTION:
In this prospective multicentre case-control study, the investigators will recruit a total of 518 patients. These will be divided into the following groups:

1. Cancer group (n=259): Patients with treatment naive, histopathology confirmed OSCC.
2. Control group (n=259): Patients who have undergone or are undergoing an upper gastrointestinal (GI) endoscopy as part of their investigation for upper GI symptoms and are found to have either - (i) A normal upper GI tract or (ii) Benign upper GI disease.

Eligible and willing participants will be asked to provide two breath samples by exhaling into single-use breath collection bags. Using a custom designed gas sampling pump, the breath VOCs will be transferred onto thermal desorption (TD) tubes at a controlled flow rate. When the participants' breath sampling is complete, room air (Blank) samples will be taken onto additional TD tubes using the same process.

Once collected, the TD tubes will be transported to Imperial College London (The Hanna lab), where they will be analysed.

ELIGIBILITY:
Inclusion Criteria: Participants with all the following characteristics will be eligible for inclusion in the study:

1. Cancer cohort (n=259): Patients with treatment naïve, histopathology confirmed OSCC.
2. Control cohort (n=259): Patients who have undergone or are undergoing an endoscopy (OGD) as part of their investigation for upper GI symptoms and are found to have either:

   * A normal upper gastrointestinal tract
   * Benign upper gastrointestinal disease

Exclusion Criteria: Participants with the following characteristics will not be eligible for inclusion in the study:

1. Received some form of treatment (chemotherapy, radiotherapy, immunotherapy, endoscopic resection, or surgery) for OSCC
2. History of another cancer in the last five years
3. Non-squamous cell oesophageal cancer
4. Barrett's oesophagus (with or without dysplasia)
5. Previous oesophageal or gastric resection
6. Unable to provide written consent or lack capacity.
7. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment naïve OSCC will be identified via the weekly multidisciplinary team (MDT) meetings (OSCC group). Patients undergoing an OGD for upper GI symptoms will be identified using the National Health Services (NHS) trust booking systems (Control group).
Sampling Method: Probability Sample
Enrollment: 518 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop a breath test for detection of OSCC | 36 months
  The investigators hypothesise that breath VOCs in OSCC are unique and different to those in non-cancer patients. Replicate breath samples will be analysed by two independent assays using different Thermal Desorption - Gas Chromatography - Time of Flight Mass Spectrometry (TD-GC-TOF-MS) instruments. One assay will use a mid-polar, and the other a polar column stationary phase for optimal determination of VOC chemical classes. The samples will then be recollected and analysed by two-dimensional (2D) TD-GC-TOF-MS for robust VOC identification. Confirming the identity of the top VOCs driving the model will provide chemical validation. Data obtained will be used to refine the model using molecular network analysis. Statistical methods will estimate the probability of OSCC as a function of measured VOCs. Calibrations and method validation will be used to assess and correct for discrimination.

SECONDARY OUTCOMES:
To evaluate the effects of known confounding variables on the target VOCs in OSCC | 36 months
  To develop this clinical triage test, the investigators will use logistic regression modelling. They will assess the linearity of relationships between OSCC risk and continuous variables and explore categorical variables and two-way interactions. Inclusion of patient characteristics (e.g., age, gender, alcohol use and smoking), clinical variables (e.g., symptoms) and VOCs in the model will be determined using a combination of statistical significance (Wald p<0.05), size of the model coefficients and clinical opinion, drawing on contemporary methods for clinical prediction rules.
  The investigators will use model reduction techniques such as the LASSO (least absolute shrinkage and selection operator) or Harrell's step-down approach to prevent over-fitting. They will also assess optimism. If there is missing data, the investigators will apply multiple imputation techniques.

CONTACTS AND LOCATIONS:
Locations (13):
- United Kingdom (13):
  - Imperial College Healthcare NHS Trust, London, Greater London
  - Hull University Teaching Hospitals NHS Trust, Cottingham, Hull
  - Cardiff and Vale University Health Board, Cardiff
  - Velindre NHS Trust, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Bedfordshire Hospitals NHS Foundation Trust, Luton
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Oxford University Hospitals NHS Trust, Oxford
  - Portsmouth Hospitals University NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No